CLINICAL TRIAL: NCT06174506
Title: The Role of hs Troponin I and NT-proBNP in Predicting Atrial Fibrillation in Patients With Permanent Pacemakers
Status: Recruiting | Type: Observational
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Linh Ha Khanh Duong, Duong Ha Khanh Linh, University of Medicine and Pharmacy at Ho Chi Minh City
Other Study IDs: 806/HDDD-DHYD
Record Dates: First submitted 2023-11-30; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood samples will be drawn from fasting participants. The blood then will be promptly processed, and serum or plasma will be used for quantification of hs Troponin I or NT-proBNP.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with pacemakers without atrial fibrillation at the beginning or in history: Patients with pacemakers without atrial fibrillation at the beginning or in history.
  Patients are adults over 18 years old.

SUMMARY:
The goal of this clinical trial is to answer the research question whether hs Troponin I and NT-proBNP have a role in detecting atrial fibrillation in patients with pacemakers.

Objectives of the study:

1. To survey some risk factors for atrial fibrillation in patients with permanent pacemakers.
2. To determine the role of hs Troponin I and NT-proBNP in predicting new-onset atrial fibrillation within follow-up time.
3. To build a model to predict the prognosis of atrial fibrillation based on the detected subclinical markers related to atrial fibrillation and classic cardiovascular risk factors.

DETAILED DESCRIPTION:
Information about age, gender, BMI, medical history, tests to evaluate liver function, kidney function, dyslipidemia, results of echocardiography, ECG, and chest X-ray will be collected from medical records and clinical examination.

The hs troponin I and NT-proBNP tests will be performed before the patient has a pacemaker.

The two tests above will be paid by research team. Patients do not have to pay for these tests.

Atrial fibrillation will be determined through ECG, holter ECG and pacemaker data.

Time to follow up patients in the study: According to the patient's follow-up visits after pacemaker placement: 1 month, 3 months, 6 months, then every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient is an adult (≥ 18 years old or older)
* There is indication for permanent pacemaker placement and patient agreement to permanent pacemaker placement
* Patient agrees to participate in the study

Exclusion Criteria:

* Patients had a diagnosis of atrial fibrillation in their past history or atrial fibrillation is discovered at the time of participating in the study
* Severe patients, at risk of death
* Pregnant
* The patient is indicated for surgery
* Patients with eGFR ≤ 30 mL/min/1.73m2
* The patient has a serious infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from the Arrhythmia Treatment Department of Cho Ray Hospital during the study period.
  Adult patients with indications for pacemaker placement, agree to participate in the study, meet the inclusion criteria and do not have the exclusion criteria will be selected for the study.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation | through study completion, an average of 2 year
  Symptomatic or asymptomatic AF that is documented by surface ECG. The minimum duration of an ECG tracing of AF required to establish the diagnosis of clinical AF is at least 30 seconds, or entire 12-lead ECG.

SECONDARY OUTCOMES:
Atrial high-rate episodes (AHRE) | through study completion, an average of 2 year
  AHRE - events fulfilling programmed or specified criteria for AHRE that are detected by CIEDs with an atrial lead allowing automated continuous monitoring of atrial rhythm and tracings storage. CIED-recorded AHRE need to be visually inspected because some AHRE may be electrical artefacts/false positives.
Subclinical AF | through study completion, an average of 2 year
  Subclinical AF includes AHRE confirmed to be AF, AFL, or an AT, or AF episodes detected by insertable cardiac monitor or wearable monitor and confirmed by visually reviewed intracardiac electrograms or ECG-recorded rhythm.

CONTACTS AND LOCATIONS:
Overall Officials: Linh HK Duong, Master, Principal Investigator — Cho Ray Hospital
Locations (1):
- Cho Ray Hospital, Ho Chi Minh City, None Selected, Vietnam

IPD SHARING:
Plan to Share IPD: No